CLINICAL TRIAL: NCT06691607
Title: The Role of Neutrophil Gelatinase Associated Lipocalin in Early Detection of Acute Kidney Injury and Prediction of Patient Outcome in Critically Ill Patients; a Prospective, Observational, Non-randomized Study
Brief Title: NGAL in Prediction of AKI and Patient Outcomes
Acronym: NGAL AKI
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fawzy Abbas Badawy, Assistant professor of Anesthesia, Sohag University
Other Study IDs: Soh-Med-23-01-31
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: To Determine If Blood Level (NGAL) Could Accurately Early Detect Acute Renal Damage in All Patients Requiring Critical Care
Keywords: Critically ill, neutrophil gelatinase-associated lipocalin, acute kidney injury.
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: Group A progressed to AKI
  Interventions: Other: Serum NGAL level
- Group B: Group B did not progress to AKI
  Interventions: Other: Serum NGAL level

INTERVENTIONS:
Other: Serum NGAL level — serum NGAL level

SUMMARY:
This single-center prospective non-randomized observational research included 120 critically ill persons, at Sohag University hospital's critical care unit. NGAL serum level was assessed at admission to the intensive care unit (NGAL1) and 24 hours after first sample (NGAL2). Cases were categorized into two groups depending on their progression or not to AKI, group A or group B respectively during their intensive care unit stay. Serum NGAL1 and NGAL2 concentrations were compared in relation to development of AKI (group A) or not (group B), need for RRT or not and in relation to mortality.

DETAILED DESCRIPTION:
Introduction A sudden and prolonged decline in renal function is defined as acute kidney injury (AKI). (1) Frequency of acute kidney injury is ranged from 30% to 67% of critically ill patient.(2,3). Nowadays the main marker used for diagnosis of AKI is serum creatinine which is functional marker, the change in its serum level may be delayed that delay diagnosis and management and may worsen outcome.(4) Within 1-4 hours following ischemic renal insult, NGAL has been shown to be detectable in the serum and urine, but until nowadays it has no clinical usage.(5, 6).

Patients and methods:

This single-center prospective non-randomized observational research has been performed on 120 cases, admitted to the critical care unit of the Sohag University Hospital between April 2020 and June 2022. A written and informed agreement was obtained from each patient or his first-degree guardian after clearance by the Sohag Faculty of Medicine's Ethics and Research Committee under IRB Registration Number: Soh-Med-23-01-31.

Inclusion criteria: All severely sick ICU patients older than 18 years old were included in the study.

Exclusion criteria: Patients with known chronic renal disease, those receiving hemodialysis, those with transplanted kidney, those with known kidney cancer, and patients who were just released from the ICU.

Methods: All included patients were subjected to the following: History taking, demographic data (age and gender), full medical history including co-morbid conditions (Chronic liver illness, ischemic heart disease, hypertension, and diabetes mellitus), medications, smoking status, previous surgeries, duration of hospital stay before ICU admission and infections including pneumonia, urinary tract infection, gastrointestinal tract, blood stream related infections or any wound infection. Complete clinical examination including BP, heart rate and O2 saturation, Glasgow coma scale (GCS), mean arterial pressure (MAP), temperature, respiration rate, oxygen saturation, presence or lack of lower limb edema, ascites and bed sores and measurement of urine output immediately on admission and every 6 hour. NGAL was measured utilizing an enzyme-linked immunosorbent assay (ELISA) sandwich method utilizing reagents from BT LAB. Symbol: E1719Hu. Size: 96T. Serum level of creatinine was measured immediately on admission and every 24 hours. Routine Laboratory investigations: Renal and liver functions, complete blood count and serum K, Na, PH, PCO2, PO2 and HCO3. Also, abdominal ultrasound comment on kidney echogenicity was performed. Utilizing the RIFLE-SCr method developed by the Acute Dialysis Quality Initiative (ADQI) group (7), participants were split into two groups: group A that advanced acute kidney injury or failure during their intensive care unit stay, and group B that didn't. Patients with AKI should consider dialysis if they have any of the following conditions: volume expansion that is resistant to diuretics, hyperkalemia resistant to medical treatment, severe acid-base disturbances resistant to medical treatment, severe azotemia (BUN >80-100), and uremia.

Primary outcome measure was the capability of serum NGAL levels to identify renal damage early in all patients requiring critical care. Secondary outcome measures were detection of patient outcome either; the need to RRT or patient mortality.

Sample size calculation Sample size was calculated using Power Analysis and Sample Size software program (PASS) version 15.0.5 for windows (2017) using data published by D. Youssef et al (2013) with the ability of NGAL to early detect renal injury in all critical care patients as the primary outcome. The null hypothesis was considered as the inability of NGAL to detect renal injury in all critical care patients. Youssef et. al (8) reported the area under the ROC curve of NGAL to early detection of AKI to be 0.63 with 95% confidence interval 0.50- 0.77.

Statistical analysis: Using IBM's SPSS statistics (Statistical Package for the Social Sciences) for Windows, the collected data were statistically examined (version 26). In order to ascertain if the data distribution was normal, the Shapiro-Wilk test was used. Regularly distributed continuous variables were stated as mean SD whereas categorical data and continuously distributed variables with aberrant distribution were given as median and interquartile range or number and percentage (as appropriate). The Student t test and Mann-Whitney tests were used, respectively, for continuous data with a normal distribution and those with an abnormal distribution. The chi square test was used to evaluate categorical data using the crosstabs function. There was a 95% confidence interval used for each test.

ELIGIBILITY:
Inclusion Criteria:

- All severely sick ICU patients older than 18 years old were included in the study

Exclusion Criteria:

* Patients with known chronic renal disease, those receiving hemodialysis, those with transplanted kidney, those with known kidney cancer, and patients who were just released from the ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All included patients were subjected to the following: History taking, demographic data, full medical history before ICU admission. Complete clinical examination immediately on admission. NGAL was measured by (ELISA) at admission and after 24 hours. Serum level of creatinine was measured immediately on admission and every 24 hours. Routine Laboratory investigations, abdominal ultrasound comment on kidney echogenicity was performed. Utilizing the RIFLE-SCr method, participants were split into two groups: group A that advanced acute kidney injury or failure during their intensive care unit stay, and group B that didn't. Patients with AKI should consider dialysis if they have been indicated.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
the capability of serum NGAL levels to identify renal damage early in all patients requiring critical care | through study completion, an average of 1 year
  the capability of serum NGAL levels to identify renal damage early in all patients requiring critical care

SECONDARY OUTCOMES:
detection of patient outcome either; the need to RRT or patient mortality. | through study completion, an average of 1 year
  detection of patient outcome either; the need to RRT or patient mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
no plan to participate indevidual data